CLINICAL TRIAL: NCT03644082
Title: Computerized Cognitive Training for Patients With Epilepsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems recruiting and retaining volunteer research personnel to assist with the recruitment of subjects and the study procedures
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-01830
Record Dates: First submitted 2018-08-21; First posted 2018-08-23 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epilepsy Patients (Experimental)
  Interventions: Behavioral: Luminosity Trial Memory Match; Behavioral: Luminosity Trial Memory Matrix; Behavioral: Luminosity Trial Famliar Faces; Behavioral: Luminosity Trial Brain Shift; Behavioral: Luminosity Trial Star Search; Behavioral: Luminosity Trial Word Bubbles; Behavioral: Luminosity Trial Color Match; Behavioral: Luminosity Trial Ebb and Flow; Behavioral: Luminosity TrialChalk Board Challenge; Behavioral: Luminosiuty Follow that Frog; Behavioral: Luminosity Train of Thought

INTERVENTIONS:
Behavioral: Luminosity Trial Memory Match — Working memory task that has users indicate whether the current symbol matches the one presented 2 symbols previously. As the user makes correct responses, the previous symbols reduce in contrast and fade int the background, ultimately disappearing, forcing the user to rely entirely on working memory to achieve success
Behavioral: Luminosity Trial Memory Matrix — The purpose id to remember the location of squares on a grid
Behavioral: Luminosity Trial Famliar Faces — The purpose is to create associations between visual and verbal information
Behavioral: Luminosity Trial Brain Shift — The purpose is to decide whether or not cards with numbers and letters are either even or vowels. This measures inhibition, flexibility, and monitoring response set. Also, letterfluency, category fluency, and category switching.
Behavioral: Luminosity Trial Star Search — The purpose is to visually scan several different objects and find the different object in array of pictures. This measures selective attention.
Behavioral: Luminosity Trial Word Bubbles — The purpose is to decide what suffix to use in order to complete a word whena prefix is given. The subject needs to come up with he ending of three different prefixes to complete the word.
  This task measures verbal modality, deductive reasoning, integration of multiple bits of information, and flexibility of thinking.
Behavioral: Luminosity Trial Color Match — The purpose is to identify whether colors and words match each other. This measures the ability to inhibit a dominant and automatic verbal response
Behavioral: Luminosity Trial Ebb and Flow — Identify which direction leaves are pointing or moving depending on their color.This measures inhibition of impulsive and perseverative responding, and the ability to establish and maintain instructional set.
Behavioral: Luminosity TrialChalk Board Challenge — purpose is to problem solve quantitative reasoningequationsand to decide which card is greater or if the 2 cards are equal when the math problem is solved.
Behavioral: Luminosiuty Follow that Frog — The purposeis to remember the path a red frog takes as it jump from lilypad to lily pad in a pond. This measures flexibility of thinking on a visual-motor sequencing task and working memory
Behavioral: Luminosity Train of Thought — purpose is to guide specific colored trains into corresponding colored matching houses by attending to the different tracks. This measures divided attention.

SUMMARY:
This is a study on the effectiveness of computerized cognitive training for treatment of memory disorders in patients with epilepsy. Participants will be recruited from patients referred for neuropsychological assessment through the NYU Comprehensive Epilepsy Center's inpatient and outpatient services. Individuals meeting inclusion criteria will be screened for the presence of memory disturbance (defined by results of neuropsychological testing) and lack of exposure to any previous form of computerized cognitive training. All eligible subjects will be provided with an account for Lumosity with instructions to complete training modules 5 days per week for a total of 8 consecutive weeks. Outcomes will be evaluated through changes on the neuropsychological test battery.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of epilepsy based on medical records. The records will be reviewed by the PI and the approved study personnel to confirm that a diagnosis of epilepsy has been made.
* Presence of memory disturbance, as defined by an immediate or delayed memory index score < 85 on the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
* Availability of a home computer and internet for access to the computer training program.

Exclusion Criteria:

* Full Scale IQ < 80, as assessed by an appropriate Wechsler scale (WAIS-IV or WASI-II).
* Epilepsy surgery within 8 weeks of the beginning of the trial.
* History of chronic progressive neurologic or neurodegenerative illnesses (e.g., Alzheimer's disease, multiple sclerosis, primary or metastatic malignancy). Patients with headache or migraine are not excluded.
* History of Axis I psychiatric illness with psychotic features. (e.g., schizophrenia or bipolar disorder). Patients with depression or anxiety (treated or untreated) without psychotic features are not excluded.
* Visual or auditory impairment, which precludes participation in part, or all of the testing or computer training.
* English as a first language will not be required, but participants must have either received some of their schooling in English or used English in their work for >10 years.
* Previous exposure (> one week) to Lumosity or a similar computerized training program.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Immediate Memory Index Score | 12 Months
  Score on the Repeatable Battery for the Assessment of Neuro-psychological Status (RBANS) will be used to measure immediate memory
Delayed Memory Index Score | 12 Months
  Score on the Repeatable Battery for the Assessment of Neuro-psychological Status (RBANS) will be used to measure immediate memory

CONTACTS AND LOCATIONS:
Overall Officials: William Barr, MD, Study Director — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No